CLINICAL TRIAL: NCT06242288
Title: Correlation Between Depression Scores and Serum NF-ĸB/NLRP3 Axis, Biotinidase, and HMGB After Treatment With Isotretinoin in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 659874
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): age and sex matched healthy control
- Comparative group (Active Comparator): 20 acne patients taking isotretinoin 20 mg once daily
  Interventions: Drug: ISOtretinoin 20 MG

INTERVENTIONS:
Drug: ISOtretinoin 20 MG — Isotretinoin, also known as 13-cis-retinoic acid and sold under the brand name Accutane among others, is a medication primarily used to treat severe acne
  Arms: Comparative group

SUMMARY:
Acne is a chronic inflammatory disease of the pilosebaceous unit resulting from androgen-induced increased sebum production, altered keratinization, inflammation, and bacterial colonization of hair follicles on the face, neck, chest, and back by, Cutibacterium acnes. Although all age groups can be affected, it is primarily a disease of adolescence. Treatment selection is based on disease severity, patient preference, and tolerability. Isotretinoin is drug of chioce used for moderate and severe acne. Isotretinoin results in a significant reduction in sebum production, influences comedogenesis, lowers surface and ductal c. acnes and has anti-inflammatory properties. Biotin deficiency may be caused by insufficient dietary uptake of biotin, drug- vitamin interactions and increased biotin catabolism during pregnancy and in smokers. Biotin deficiency can also be precipitated by decreased activities of biotinidase, which plays a central role in the intestinal absorption of biotin

ELIGIBILITY:
Inclusion Criteria:

Age of 19 to 35 years. Body mass index (BMI) of 18.5 to 23 kg/m2. Acne vulgaris (global acne scoring more than 18)

Exclusion Criteria:

Use of oral steroids, oral contraceptives, oral vitamin A derivatives, antibiotics, or herbal medicines that may affect the test results during the last 4 weeks.

Alcohol drinking within the last week. Smoking. Pregnancy or lactation. Judgement that physical or mental testing is not appropriate for the clinical trial.

Participation in other clinical trials that may affect this t

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
change in biotinidase level | 2 months
  change in biotinidase level

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt